CLINICAL TRIAL: NCT01009229
Title: A Reduced 11 Beta Hydroxysteroid Dehydrogenase 2 (11 Beta HSD2) Activity, a Novel Mechanism of Salt Sensitivity and Hypertension After Renal Allograft Donation?
Brief Title: A Reduced 11-b-HSD Activity, a Novel Mechanism of Salt Sensitivity and Hypertension After Renal Allograft Donation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Felix Frey, Department of Nephrology and Hypertension, University of Berne, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uehlinger-001
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Renal Failure; Renal Transplantation; Living Donors
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Dietary Supplement: Low and high salt diets

INTERVENTIONS:
Dietary Supplement: Low and high salt diets — High salt diet: 150mmol/d Low salt diet: 30mmol/d
  Other Names: NaCl

SUMMARY:
Consecutive living-kidney donor candidates (n=100) will be recruited after being accepted for donation according to official guidelines. An assessment of salt sensitivity, 11 beta HSD activity, 24 hour blood pressure, urine collection and physical exam will be performed prior nephrectomy and 14, 52, 156, 208 days post-nephrectomy.

DETAILED DESCRIPTION:
Consecutive living-kidney donor candidates (n=100) will be recruited after being accepted for donation. The assessment of salt sensitivity, 11 beta HSD activity, 24 hour blood pressure, urine collection and physical exam will be performed prior nephrectomy and 14, 52, 156, 208 days post-nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* acceptance for living kidney donation

Exclusion Criteria:

* withdrawal of consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Salt sensitivity, arterial hypertension | day 0, 14, 52, 156, 208, yearly

CONTACTS AND LOCATIONS:
Overall Officials: Felix J Frey, Prof, Principal Investigator — University of Berne
Locations (1):
- Department of nephrology and hypertension, Universitiy of Bern, Bern, Canton of Bern, Switzerland